CLINICAL TRIAL: NCT04570020
Title: Clinical Trial of OCT-based Scleral Lens Fitting With Wide-Field OCT
Brief Title: Scleral Lens Fitting Using Wide-Field OCT
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, David Huang, Peterson Professor of Ophthalmology & Professor of Biomedical Engineering, Oregon Health and Science University
Other Study IDs: 6612-SCLERAL LENS; R01EY028755 (NIH)
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus; Irregular; Contour of Cornea
Keywords: Keratoconus (KCN); Irregular Cornea; Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Clinically-Selected Scleral Lens: The clinically-selected lens is based on slit lamp assessment. This lens will be compared against an OCT-selected lens.
- OCT-Selected Scleral Lens: The OCT-selected lens is based on OCT measurements. This lens will be compared against a clinically-selected lens.

SUMMARY:
The purpose of this study is to see if OCT technology can optimize scleral contact lens fittings. Subjects with keratoconus, post-penetrating keratoplasty (PK), post-LASIK ectasia, post-radial keratotomy (RK), or a variety of anterior surface disorders requiring scleral lens fittings will be considered for enrollment. For each study eye, a clinically-selected scleral lens fit will be compared against an OCT-selected lens fit. The quality of each lens fit will be determined by flourescein exam at the slit lamp. Apical clearance, limbal clearance, conjunctival compression, and lens edge lift will be assessed. A lens that satisfies all four criteria will be considered satisfactory.

ELIGIBILITY:
Inclusion Criteria:

* Eyes requiring fit for scleral lenses for KCN, post-PK, post-RK, post-LASIK ectasia, or various anterior surface disorders

Exclusion Criteria:

* Inability to maintain stable fixation for OCT imaging
* Inability to commit to required visits to complete the study
* Eyes with concurrent retinal diseases, glaucoma, or other eye conditions that may limit visual outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects meeting the eye criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Apical Clearance | 5 years
  Apical clearance of each lens (whether clinically-selected or OCT-selected) will be graded as "acceptable," "too high," or "too low."
Limbal Clearance | 5 years
  Limbal clearance of each lens (whether clinically-selected or OCT-selected) will be graded as "acceptable," "too much," or "too little."
Conjunctival Compression | 5 years
  Conjunctival compression of each lens (whether clinically-selected or OCT-selected) will be graded as "acceptable" or "excessive."
Lens Edge Lift | 5 years
  Lens edge lift for each lens (whether clinically-selected or OCT-selected) will be graded as "acceptable" or "excessive."

CONTACTS AND LOCATIONS:
Overall Officials: David Huang, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Casey Eye Institute, Portland, Oregon, United States